CLINICAL TRIAL: NCT04599569
Title: Influence of Renal Replacement TherApy on Indirect Calorimetry: a Prospective Observational Study
Brief Title: Influence of Renal Replacement TherApy on Indirect Calorimetry
Acronym: IRATIC
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Sirak Petros, MD, Professor, University of Leipzig
Other Study IDs: IRATIC-2020
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Acute Renal Failure; Mechanical Ventilation
Keywords: indirect calorimetry; energy expenditure; carbon dioxide elimination; renal replacement therapy; respiratory quotient
MeSH Terms: conditions — Acute Kidney Injury | interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: indirect calorimetry — indirect calorimetry with and without renal replacement therapy

SUMMARY:
Renal replacement therapy may affect carbon dioxide elimination, which may theoretically influence measurement of energy expenditure by means of indirect calorimetry. However, available clinical studies are noct conclusive on this issue. This observational study aims to investigate the effect of renal replacement therapy on indirect calorimetry in critically ill mechanically ventilated patients.

DETAILED DESCRIPTION:
Optimal Nutrition of the critically ill is still a clinical challenge. Current guidelines recommend that measurement of energy expenditure using indirect calorimetry should be favoured in critically ill patients. The technique is based on measurement of oxygen consumption and carbon dioxide elimination. Experimental studies have reported on carbon dioxide elimination via renal replacement therapy. Since acute kidney injury with requirement for renal replacement therapy (RRT) is common in the intensive care unit, the significance of carbon dioxide elimination via the dialyser should be clarified. However, available evidence from clinical studies is contradictory, one reason being the heterogenous study design.

In this prospective observational study on critically ill mechanically ventilated medical patients requiring RRT, indirect calorimetry (IC) will be conducted twice on the same day with and without RRT: either immediately before commencement of RRT followed by a second IC with RRT after an RRT run time of an hour, or immediately before the end of an RRT session followed by a second IC an hour after the termination of RRT.

ELIGIBILITY:
Inclusion Criteria:

* simultaneous requirement for mechanical ventilation and renal replacement therapy
* informed consent

Exclusion Criteria:

* age <18 years
* requirement for therapeutic hypothermia
* serum lactate >4 mmol/l
* requirement for inspiratory oxygen fraction >0.6 and positive end-expiratory pressure >12 mbar
* leak in the ventilator circuit (e.g. due to a chest tube)
* requirement for extracorporeal circulatory support
* refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill mechanically ventilated medical patients requiring renal replacement therapy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
energy expenditure | 60 minutes
  energy expenditure in kcal/d

SECONDARY OUTCOMES:
Carbon dioxide elimination | 60 minutes
  Carbon dioxide elimination in ml/min
respiratory quotient | 60 minutes
  respiratory Quotient, defined as the Ratio of Carbon dioxide elimination to Oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: Sirak Petros, MD, Principal Investigator — University of Leipzig
Locations (1):
- University Hospital of Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Knoll A, Petros S, Pasieka B, Weidhase L. Influence of kidney replacement therapy on indirect calorimetry in critically ill patients. Eur J Clin Nutr. 2025 Nov;79(11):1144-1148. doi: 10.1038/s41430-025-01643-9. Epub 2025 Jul 30. PMID 40739037